CLINICAL TRIAL: NCT04873284
Title: Comparative Study of Fosaprepitant and Aprepitant for the Prevention of Chemotherapy-induced Nausea and Vomiting in Pediatric Cancer Patients：A Superiority Design, Phase III Randomized Trial
Brief Title: Comparative Study of Fosaprepitant and Aprepitant for the Prevention of Chemotherapy-induced Nausea and Vomiting in Pediatric Caner Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fosaprepitant and aprepitant
Record Dates: First submitted 2021-04-22; First posted 2021-05-05 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Chemotherapy Induced Nausea and Vomiting; Pediatric Cancer Patients
Keywords: fosaprepitant; aprepitant; pediatric cancer; vomiting; efficacy; safety
MeSH Terms: conditions — Vomiting; Neoplasms | interventions — fosaprepitant; Aprepitant; Granisetron; Dexamethasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fosaprepitant (Experimental): Patients received intravenous Granisetron plus dexamethasone followed by fosaprepitant infusion
  Interventions: Drug: fosaprepitant; Drug: Granisetron plus dexamethasone
- Aprepitant (Experimental): Patients received intravenous Granisetron plus dexamethasone followed by oral aprepitant
  Interventions: Drug: aprepitant; Drug: Granisetron plus dexamethasone

INTERVENTIONS:
Drug: fosaprepitant — Granisetron+dexamethasone: granisetron:40mcg/kg, IV ; dexamethasone : S<0.6m2, 2 mg/dose, q12h IV/PO; S>0.6m2, 4 mg/dose, q12h , IV/PO. When used with fosaprepitant, dexamethasone dose was halved.
  Fosaprepitant: 4 mg/kg IV
  Arms: Fosaprepitant
Drug: aprepitant — Granisetron+dexamethasone: granisetron:40mcg/kg, IV ; dexamethasone : S<0.6m2, 2 mg/dose, q12h IV/PO; S>0.6m2, 4 mg/dose, q12h , IV/PO. When used with aprepitant, dexamethasone dose was halved.
  Oral aprepitant: D1：Powder for suspension 3.0 mg/kg (up to 125 mg),D2，D3：Powder for suspension 2.0 mg/kg (up to 80 mg).
  Arms: Aprepitant
Drug: Granisetron plus dexamethasone — Granisetron+dexamethasone: granisetron:40mcg/kg, IV ; dexamethasone : S<0.6m2, 2 mg/dose, q12h IV/PO; S>0.6m2, 4 mg/dose, q12h , IV/PO.

SUMMARY:
Children aged 2-12 years scheduled to receive moderately or highly emetogenic chemotherapy were randomly assigned to arm-A (fosaprepitant) or arm-B (aprepitant). Children recruited to arm-A received intravenous granisetron plus dexamethasone followed by fosaprepitant infusion. Children recruited to arm-B received the same drugs as those given to children in arm-A, except that fosaprepitant was substituted with aprepitant. Granisetron and dexamethasone were given continuously until 48 hours after completion of chemotherapy. The primary end point of the study was to determine the proportion of patients who achieved a CR, defined as no vomiting, no retching, and no use of rescue medication, the proportion of patients who achieved a CR during the acute phase (0-24 hours) after administration of the last dose of chemotherapy. Secondary end points were the proportion of patients who achieved a CR during the 24-120 hours (delayed phase) and overall after administration of the last dose of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

children aged 2-12 years at the time of study entry with documented cancer scheduled to receive MEC or HEC (more than 30% emetogenic potential) with Karnofsky score of 60 or more (for patients aged greater than 10 years) or Lansky play performance score of 60 or more (for patients aged 10 years or less) predicted life expectancy of at least 3 months; and written informed consent provided by parent or guardian

Exclusion Criteria:

vomiting 24 hours before treatment day 1 known history of QT prolongation or allergic reaction to any of the study drugs symptomatic primary or metastatic CNS malignancy causing nausea or vomiting patients who received radiation therapy to the abdomen or pelvis in the week before treatment; active infection or any uncontrolled concurrent illness except for malignancy abnormal laboratory values at screening (peripheral absolute neutrophil count <1000 cells per μL, platelet count <100 000 cells per μL; alanine amino transferase or aspartate aminotransferase >5 times of the upper limit of normal for age, bilirubin or serum creatinine >1.5 times of the upper limit of normal for age) initiation of systemic corticosteroids within 72 hours before study drug administration or as part of the chemotherapy regimen; benzodiazepines or opioids initiated within 48 hours before treatment, except for single doses of triazolam, temazepam, or midazolam use of antiemetics within 48 hours of treatment use of CYP3A4 substrates or inhibitors within 7 days or CYP3A4 inducers within 30 days of treatment

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-12-25 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete Remission rates in the acute phases | up to 6 months
  The primary end point was complete remission rates in the acute phase. Complete Remission was defined as no vomiting, no retching, and no use of rescue medication

SECONDARY OUTCOMES:
Complete Remission rates in the delayed and overall phases | up to 6 months
  Complete Remission rates in the delayed and overall phases
Adverse events reported in study patients | up to 6 months
  All of the adverse reactions of aprepitant and fosaprepitant during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jin Gao, Study Director — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flank J, Robinson PD, Holdsworth M, Phillips R, Portwine C, Gibson P, Maan C, Stefin N, Sung L, Dupuis LL. Guideline for the Treatment of Breakthrough and the Prevention of Refractory Chemotherapy-Induced Nausea and Vomiting in Children With Cancer. Pediatr Blood Cancer. 2016 Jul;63(7):1144-51. doi: 10.1002/pbc.25955. Epub 2016 Mar 9. PMID 26960036
- [Background] Weinstein C, Jordan K, Green SA, Camacho E, Khanani S, Beckford-Brathwaite E, Vallejos W, Liang LW, Noga SJ, Rapoport BL. Single-dose fosaprepitant for the prevention of chemotherapy-induced nausea and vomiting associated with moderately emetogenic chemotherapy: results of a randomized, double-blind phase III trial. Ann Oncol. 2016 Jan;27(1):172-8. doi: 10.1093/annonc/mdv482. Epub 2015 Oct 8. PMID 26449391
- [Background] Radhakrishnan V, Joshi A, Ramamoorthy J, Rajaraman S, Ganesan P, Ganesan TS, Dhanushkodi M, Sagar TG. Intravenous fosaprepitant for the prevention of chemotherapy-induced vomiting in children: A double-blind, placebo-controlled, phase III randomized trial. Pediatr Blood Cancer. 2019 Mar;66(3):e27551. doi: 10.1002/pbc.27551. Epub 2018 Nov 13. PMID 30426714
- [Background] Mora J, Valero M, DiCristina C, Jin M, Chain A, Bickham K. Pharmacokinetics/pharmacodynamics, safety, and tolerability of fosaprepitant for the prevention of chemotherapy-induced nausea and vomiting in pediatric cancer patients. Pediatr Blood Cancer. 2019 Jun;66(6):e27690. doi: 10.1002/pbc.27690. Epub 2019 Mar 21. PMID 30900392
- [Background] Dupuis LL, Boodhan S, Holdsworth M, Robinson PD, Hain R, Portwine C, O'Shaughnessy E, Sung L; Pediatric Oncology Group of Ontario. Guideline for the prevention of acute nausea and vomiting due to antineoplastic medication in pediatric cancer patients. Pediatr Blood Cancer. 2013 Jul;60(7):1073-82. doi: 10.1002/pbc.24508. Epub 2013 Mar 19. PMID 23512831
- [Derived] Yu LT, Wang Z, Han YL, Zhou F, Wagner LM, Zhang SG, Li ZL, Gao YJ. Comparison of oral aprepitant and intravenous fosaprepitant for prevention of chemotherapy-induced nausea and vomiting in pediatric oncology patients: a randomized phase III trial. Transl Pediatr. 2024 Jan 29;13(1):110-118. doi: 10.21037/tp-23-598. Epub 2024 Jan 12. PMID 38323173